CLINICAL TRIAL: NCT03174145
Title: Validation Study to Investigate the Effect of a New Treatment in Patients With Osteoarthritic Pain of Knee or Hip
Brief Title: Validation Study to Investigate the Effect of a New Treatment in Patients With Osteoarthritic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tools4Patient (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: T1010-01
Record Dates: First submitted 2017-05-29; First posted 2017-06-02 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Pharmacogenomic Testing; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator)
  Interventions: Behavioral: Positive behaviour; Drug: T4P1010 administration; Genetic: Pharmacogenetic; Other: Questionnaires and diary completion
- Control group (Sham Comparator)
  Interventions: Genetic: Pharmacogenetic; Other: Questionnaires and diary completion

INTERVENTIONS:
Behavioral: Positive behaviour — Information about T4P1010 treatment
  Arms: Active group
Drug: T4P1010 administration — Provide treatment to be taken twice a day between Visit 2 and Visit 5 as add-on therapy to patient's regular analgesic treatment
  Arms: Active group
Genetic: Pharmacogenetic — Blood sample of 10 millilitres maximum
Other: Questionnaires and diary completion — Personality, pain and disease questionnaires completion during the study Diary completion between Visit 1 and Visit 5

SUMMARY:
The purpose of this clinical trial conducted in patients suffering from chronic pain is to study the relationship between individual patients' profile and their analgesic response

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of at least 18 years of age.
2. Osteoarthritis (OA) of knee or hip diagnosed since at least 6 months.
3. Affiliated with national welfare.
4. Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
5. Have given written informed consent approved by the relevant Ethics Committee governing the study sites.
6. Pain scores reported during the baseline period preceding randomization with a mean APS on the last 14 reported values before Visit 2 between 3.6 and 8.4 inclusive and to have completed at least 2/3 of each pain score in their diary between Visit 1 and Visit 2.
7. Patient with a unilateral or bilateral OA of the knee or hip diagnosed according to the American College of Rheumatology (ACR) criteria based on clinical and radiographic evidence (Altman et al., 1986) (in case of bilateral OA or OA of both knee and hip, the joint to consider should be the most affected one). The clinical diagnosis of OA will be confirmed by the ACR clinical criteria and medical imaging criteria for classification of OA of the knee or hip based upon the following criteria:

   1. Knee or hip pain as an average at least half of the time for the last 3 months before screening visit.
   2. OA of the knee, at least 1 of the following 3 conditions:

   i. age > 50, ii. morning stiffness <30 minutes, iii. crepitus on active motion and osteophytes.

   OA of the hip, at least 2 of the following 3 conditions:

   i. erythrocyte sedimentation rate < 20mm/hour, ii. femoral and/or acetabular osteophytes, iii. joint space narrowing (superior, axial, and/or medial). c. Kellgren and Lawrence grade > 1 as assessed by a recent medical imaging of the referred joint to confirm the diagnosis. If no imaging available, a new anterior- posterior view will be obtained and reviewed by Investigator or his/her delegate(s) to verify that the patient meets the disease diagnostic criteria.

   Exclusion Criteria:
8. Change in the " regular analgesic therapy " or introduction of a " regular analgesic therapy " (if none beforehand) for OA in the last 4 weeks prior to Visit 1 or during the study.
9. Invariable pain scores reported between Visit 1 and Visit 2 (systematically the same minimum score reported all along, the same mean score reported all along and the same maximum score reported all along).
10. Have initiated (or plan to initiate) a program (or modify an existing program in frequency and/or intensity) of physiotherapy or behavioral therapy such as pain self-management, hypnosis, sophrology, meditation program within 2 weeks prior to Visit 1 or during the study.
11. Pregnant, breastfeeding, or willing to be pregnant during the study.
12. Patients with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the patient's participation in the study.
13. Uncontrolled epilepsy.
14. Any current primary psychiatric condition, including depression or personality disorders (such as Axe II of Diagnostic and Statistical Manual of Mental Disorders (DSM-V); personality disorders and mental retardation).
15. Alcohol dependence or regular use of known drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and phencyclidine).
16. Any other relevant medical disorder/acute disease state/pain condition like fibromyalgia, lumbalgia, generalized OA judged by the Investigator as likely to interfere with the trial or represent a risk for the patient.
17. Any close relationship with the Investigators or the Sponsor (i.e. belonging to immediate family or subordination link).
18. Under legal protection, according to the national law.
19. Having completed or withdrawn from this study or any study investigating T4P1001.
20. Patient currently enrolled in a clinical trial involving use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study, or in an exclusion period according to the national law.
21. Have planned total knee or hip replacement intervention of the referred joint.
22. Reduced mobility due to OA (use of lower extremity assistive devices other than a cane or a knee sleeve such as crutches or walker or a knee brace or a "shoe lift" in relation to OA is not allowed).
23. Use or plan to use systemic corticosteroids 4 weeks prior to Visit 1 or during the study; Intra-muscular corticosteroid injections or Intra-articular injection of steroids into the referred knee/hip within 3 months before Visit 1 or during the study; Intra-articular injection of corticosteroids into any other sites than the referred knee/hip within 4 weeks prior to Visit 1 or during the study (corticosteroids in topical use are allowed).
24. Have used viscosupplementation or intra articular injection of hyaluronic acid in the referred joint within 3 months prior to Visit 1 or plan to use during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Patient's change from baseline of pain severity, as measured by the weekly means of the daily Average Pain Score (APS) in the last 24 hours during a 12-week treatment therapy period | Time zero equals baseline (Day-28) up to Day 85
  11-point Numeric Rating Scale (NRS)

SECONDARY OUTCOMES:
Patient's change from baseline of pain severity as measured by the weekly means of the worst pain score (WPS) in the last 24 hours | Time zero equals baseline (Day-28) up to Day 85
  11-point NRS
Patient's change from baseline of pain severity as measured by the weekly means of the least pain score (LPS) in the last 24 hours | Time zero equals baseline (Day-28) up to Day 85
  11-point NRS
Patient's change from baseline of condition as measured by the western Ontario and McMaster universities arthritis index (WOMAC) | From baseline (Day-28) up to Day 85
  Scales
Patient's change from baseline of pain severity as measured by the brief pain inventory (BPI) | From baseline (Day-28) up to Day 85
  Scales
Patient's change from baseline of Investigator and Patient Global Assessment of Changes (IGAC and PGAC) | From baseline (Day-28) up to Day 85
  11-point NRS
Cronbach alpha assessment of MPSQ | Day 1 and Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pereira, Study Director — Tools4Patient
Locations (6):
- CHU Liège, Médecine de l'appareil locomoteur, Liège, Belgium
- France (3):
  - Eurofins Optimed, Gières
  - Hopital Saint Antoine AP-HP Rhumatologie, Paris
  - Hopital Cochin AP-HP Evaluation et traitement de la Douleur, Paris
- United Kingdom (2):
  - Mac Clinical Research, Cannock
  - Mac Clinical Research, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trial Results published on EU Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2017-001028-23/results